CLINICAL TRIAL: NCT03769974
Title: Evaluation of Motor Learning on a Sequence of Manual Motor Gestures of Increasing Complexity Through the Action Observation Training and Motor Imagery: a Randomized Controlled Trial.
Brief Title: Evaluation of Motor Learning on a Sequence of Manual Motor Gestures of Increasing Complexity Through the Mental Practise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Motor Activity
Keywords: motor imagery; action observation; motor learning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An independent blind assessor will perform the measurements and recorded the data. Finally, the participants will also be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery (Experimental): A group of healthy subjects who meet the inclusion and exclusion criteria established for the study to which a first-person kinesthetic motor imagery training will be conducted on a sequence of manual motor gestures of increasing complexity for four consecutive days. The tasks of motor imagery will be 2 series of 30 seconds for each of the 12 manual positions to remember
  Interventions: Behavioral: Motor imagery
- Action observation (Experimental): A group of healthy subjects who meet the inclusion and exclusion criteria established for the study to which a first-personaction observation training will be conducted on a sequence of manual motor gestures of increasing complexity for four consecutive days. The tasks of action observation will be 2 series of 30 seconds for each of the 12 manual positions to remember in video format.
  Interventions: Behavioral: Action observation
- Placebo group (Placebo Comparator): A group of healthy subjects who meet the inclusion and exclusion criteria established for the study to which an imagery training and placebo observation, inspired by a rural landscape, will be given for four consecutive days. This group will carry out the observation and imagination of a landscape during 2 series of 30 seconds for each manual motor sequence to remember.
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Motor imagery — Two series of 30 seconds training of motor imagery in each manual engine gesture
  Arms: Motor imagery
Behavioral: Action observation — Two series of 30 seconds training of action observation training in video format in each manual engine gesture
  Arms: Action observation
Behavioral: Placebo intervention — Two series of 30 seconds of observation and imagination of a landscape during for each manual motor sequence
  Arms: Placebo group

SUMMARY:
The main objective of this research is to evaluate and quantify successes and errors, as well as execution time, in a sequence of manual motor gestures of increasing complexity through mental practice training (observation of actions and motor imagery).

DETAILED DESCRIPTION:
The motor programs stored in the procedural memory systems allow the generation of motor mental images without the need for an external stimulus, although it has been demonstrated that providing visual information, prior to a task of imagination, facilitates it and causes a greater neurophysiological activity than if it were done in an isolated manner. Some studies have shown that in the short term, in complex motor tasks of foot and hand in a coordinated manner, the action observation training provokes a greater motor learning compared to the motor imagery strategy.

However, these studies have only assessed short-term memory immediately after the intervention. No study has so far evaluated these improvements in motor learning through action observation training and motor imagery on consecutive days, nor has it been evaluated with short to medium-term follow-up.

It is therefore that there is a lack in the current scientific literature regarding which isolated method, without physical practice, of mental practice on motor learning is the most effective when exposed both on consecutive days, as well as to short-medium-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no pain subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material. Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-07-10 (Estimated); Study Completion 2019-08-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of successes in finger positions | changes in the success rates at the end of the intervention, 7 days, 1 month and 4 months after the end of the intervention
  During the measurements, the percentage of hits and errors achieved in each hand position in each of the manual engine sequences will be evaluated.
Execution time | changes in the success rates at the end of the intervention, 7 days, 1 month and 4 months after the end of the intervention
  During each measurement, the time required for each participant to place their hands will be recorded.

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Pre-intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with MIQ-R Questionnaire. MIQ-R has 4 movements repeated in two subscales, a visual and a kinaesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. A modification was made in the MIQ-R. Items 2 and 5, in which a small jump is made, were changed by standing on tiptoe. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale.
Mental Chronometry | Pre-intervention
  Mental chronometry evaluation was also used to measure the subject's motor imagery ability. Using a stopwatch, the time spent for performing each MIQ-R task was recorded. Time recorded corresponds to the interval between the command to start the task, given by the evaluator, and the verbal response of conclusion of the task, given by the subject. Mental chronometry is a reliable behavioral task that has previously been employed to collect an objective measure of MI ability
The degree of physical activity | Pre-intervention
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive
Laterality task | Pre-intervention
  With the task of recognition of the hand's laterality, two aspects will be evaluated: first, the precision (percentage of correct answers) of the discrimination of the laterality which is the capacity to recognize if a part of the body belongs to the right or left hemicorpse and second, the response time that the participants use in the task of discrimination or cognitive judgment. The app designed and developed by the NOI group will be used.
Memory Operation Questionnaire | Pre-intervention
  The allows a cognitive evaluation of everyday memory failures. The questionnaire contains four subscales: daily memory, text recall, past memories and mnemonic strategies. The memory functioning questionnaire has adequate psychometric properties of validity and reliability obtained. An acceptable internal consistency was obtained, with a Cronbach alpha coefficient of the total scale of 0.818 memory operation questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No